CLINICAL TRIAL: NCT06324123
Title: Observational Study Aimed at Evaluating the Trend of Neuropathic Pain Through the Reduction of the NRS Questionnaire Score in Patients Treated With PEACETIL
Brief Title: Observational Study Aimed at Evaluating the Trend of Neuropathic Pain
Acronym: NEURATIL
Status: Completed | Type: Observational
Sponsor: Istituto Auxologico Italiano (Other)
Responsible Party: Sponsor
Other Study IDs: 23C304
Record Dates: First submitted 2024-03-06; First posted 2024-03-21 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Neuropathic Pain
Keywords: Neuropathic Pain
MeSH Terms: conditions — Neuralgia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with neuropathic pain: Patients with acute or chronic neuropathic pain
  Interventions: Other: Peacetil

INTERVENTIONS:
Other: Peacetil — Nutraceutical supplement Peacetil for a period of 2 months

SUMMARY:
The present study aims to evaluate the trend of neuropathic pain in patients treated with Peacetil for a period of two months.

Neuropathic pain will me assessed through the Numeric Rating Scale (NRS) questionnaire score.

ELIGIBILITY:
Inclusion Criteria:

* Patients with new or recent diagnosis of acute or chronic neuropathic pain in which the clinician decides to introduce treatment with PEACETIL according to common clinical practice, belonging to one of the following categories:
* Dysmetabolic polyneuropathy (e.g. diabetic neuropathy),
* Chemotherapy treatment neuropathy,
* Compressive mononeuropathy,
* Radiculopathy,
* Postherpetic and non-postherpetic trigeminal neuralgia;

  * The patient must be able to understand the informed consent of the study;
  * Must adhere to the procedures established by the study;
  * DN4 score >4 at T0 (month 0);

Exclusion Criteria:

* Neurological disorders confounding the primary objective;
* Clinical condition which during the observational study requires the introduction or modification of the dosage of drugs which are also indicated for the treatment of acute or chronic pain
* Introduction or modification of the dosage of drugs used to treat acute and chronic neuropathic pain (including other nutraceuticals) from 30 days before the start of the study until the end of the study.
* Presence of unstable psychiatric illness, cognitive impairment, dementia, or substance abuse that would compromise the participant's ability to provide informed consent, as judged by the investigator;
* Clinically significant unstable medical condition (e.g., cardiovascular instability, systemic infection, untreated thyroid dysfunction, serious laboratory test abnormality, or clinically significant ECG changes) that would pose a risk to the participant if they were to participate in the study, in the judgment of the 'investigator.

Ages: 18 Years to 82 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Monitoring of the reduction of neuropathic pain after 1 month and after 2 months of treatment with the nutraceutical PEACETIL, introduced according to clinical practice, and 1 month after the end of treatment.
  Evaluation of the pain scale upon signing of the consent, after 1 month, after two months of treatment and after 1 month from the suspension of PEACETIL using the following questionnaires:
  * Numerical Rating Scale (NRS);
  * Visual Rating Scale (VAS);
  * DN4 questionnaire.
Sampling Method: Probability Sample
Enrollment: 122 (Actual)
Dates: Start 2023-06-09 (Actual); Primary Completion 2024-06-20 (Actual); Study Completion 2024-06-20 (Actual)

PRIMARY OUTCOMES:
Change in neuropathic pain after two months of treatment with Peacetil | At enrollment and at two months after the start of treatment with Peacetil
  Assessed by the Numerical Rating Scale (NRS) score

SECONDARY OUTCOMES:
Change in neuropathic pain after one month of treatment with Peacetil | At enrollment and at one month after the start of treatment with Peacetil
  Assessed by the Numerical Rating Scale (NRS) score

CONTACTS AND LOCATIONS:
Locations (3):
- Italy (3):
  - Istituto Auxologico Italiano, Milan, Lombardy
  - ASST Fatebenefratelli Sacco, Milan
  - Fondazione Don Carlo Gnocchi ONLUS, Milan

IPD SHARING:
Plan to Share IPD: Undecided